CLINICAL TRIAL: NCT02156752
Title: Using Novel Behavioral Approaches to Improve Long-Term Weight Loss Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5K23KDK097143
Record Dates: First submitted 2014-05-22; First posted 2014-06-05 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ACT (Experimental): Behavioral weight loss plus techniques from Acceptance and Commitment Therapy
  Interventions: Behavioral: ACT
- SR (Active Comparator): Behavioral weight loss plus self-regulation techniques
  Interventions: Behavioral: SR
- WLO (Active Comparator): Behavioral weight loss plus cooking tips and demonstrations
  Interventions: Behavioral: WLO

INTERVENTIONS:
Behavioral: ACT — Treatment is based on Acceptance and Commitment Therapy
  Arms: ACT
Behavioral: SR — Treatment is based on Self-Regulation theory.
  Arms: SR
Behavioral: WLO — Treatment is based on cooking tips and demonstrations.
  Arms: WLO

SUMMARY:
This project is a randomized controlled trial to compare the efficacy of two interventions- one based on Acceptance and Commitment Therapy (ACT) and one based on Self-Regulation (SR)- and a control group (called weight loss only (WLO)) on 24-month weight loss outcomes. All participants will first participate in an initial 4-month standard behavioral weight loss program. Participants will be randomized into 1 of 3 groups and receive a 3-part workshop; the ACT workshop will teach ACT skills including acceptance and mindfulness techniques designed to promote behavior change and health behavior persistence consistent with one's core values. The SR program will focus on self-regulation, regular weighing, and modeling behavior on successful maintainers. The WLO group will receive a control workshop focused on cooking demonstrations and general nutrition topics.The primary outcome is weight loss at 24 months. The secondary outcome is change in psychological flexibility, a critical component of ACT interventions and a potential innovative mediating mechanism. Primary Hypothesis: At 24 months, the ACT group will show significantly greater weight loss as compared to the SR and WLO groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27.5-40
* Age 30-65

Exclusion Criteria:

* currently participating in a weight loss program
* pregnant or planning to become pregnant
* medical condition that would preclude physical activity
* terminal illness
* plans to relocate
* history of substance abuse or psychological problems that are judged by the investigators to be likely to interfere with study participation

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-07-01 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Weight | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lillis, Ph.D., Principal Investigator — Lifespan/ The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Lillis J, Dunsiger S, Thomas JG, Ross KM, Wing RR. Novel behavioral interventions to improve long-term weight loss: A randomized trial of acceptance and commitment therapy or self-regulation for weight loss maintenance. J Behav Med. 2021 Aug;44(4):527-540. doi: 10.1007/s10865-021-00215-z. Epub 2021 Mar 27. PMID 33772702
- [Derived] Lillis J, Thomas JG, Levin ME, Wing RR. Self-stigma and weight loss: The impact of fear of being stigmatized. J Health Psychol. 2020 Jun;25(7):922-930. doi: 10.1177/1359105317739101. Epub 2017 Nov 6. PMID 29105491